CLINICAL TRIAL: NCT03301831
Title: Intervention Pilot With Parents of Technology-Dependent Children
Brief Title: Resourcefulness Intervention With Parents of Technology-Dependent Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Valerie Toly, Assistant Professor- UH Research Associate, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 08-10-30; 1R15NR017302-01 (NIH)
Record Dates: First submitted 2017-09-24; First posted 2017-10-04 (Actual); Results first posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-09

CONDITIONS: Depressive Symptoms; Multiple Chronic Conditions; Family Caregivers
Keywords: Parents; Technology-Dependent Child; Resourcefulness
MeSH Terms: conditions — Depression; Multiple Chronic Conditions

STUDY DESIGN:
Intervention Model Description: 2-arm RCT with participants randomized to either the intervention or attention control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resourcefulness Training Intervention (Experimental): The intervention arm will receive an intervention that includes: a face-to-face session for teaching social (help-seeking) and personal (self-help) resourcefulness skills; ongoing access to video vignettes of caregivers of technology-dependent children describing resourcefulness skill application in daily life; 4 weeks of skills' reinforcement using daily journal writing; weekly phone calls for the first 4 weeks; and booster sessions at 2 and 4 months post enrollment.
  Interventions: Behavioral: Resourcefulness Training
- Attention Control (No Intervention): The Attention Control arm will receive weekly phone calls for the first 4 weeks and at 2 and 4 months post enrollment plus any usual care.

INTERVENTIONS:
Behavioral: Resourcefulness Training — Cognitive-behavioral intervention that includes personal and social resourcefulness skills.
  Arms: Resourcefulness Training Intervention

SUMMARY:
Technology-dependent children, those who live at home but rely on medical equipment such as mechanical ventilation or feeding tubes, require complex care for their chronic condition. Parents usually provide a majority of their care and are often overwhelmed by the caregiving demands resulting in deterioration of their own mental and physical health. The goal of this 2-arm (intervention vs. attention control) RCT is to test a cognitive-behavioral Resourcefulness Training intervention that includes teaching social (help-seeking) and personal (self-help) resourcefulness skills; ongoing access to video vignettes of caregivers of technology-dependent children describing resourcefulness skill application in daily life; 4 weeks of skills' reinforcement using daily journal writing; weekly phone calls for the first 4 weeks; and booster sessions at 2 and 4 months post enrollment. The intervention is proposed to improve these caregivers' mental and physical health outcomes and family functioning outcomes while they continue to provide vital care for these vulnerable children.

DETAILED DESCRIPTION:
Technology-dependent children, those who rely on medical equipment such as mechanical ventilation or feeding tubes for daily care at home, are among the sickest and most vulnerable subset of children with complex chronic conditions. An estimated 600,000 children in the United States are technology dependent and live at home, and are cared for primarily by their parents. These parents report greater levels of depressive symptoms and stress than other caregiver groups. In addition, these caregivers report poor psychological and physical health that compromise their caregiving capacity and increase their use of emergency rooms (ER) for their children's care needs. Despite these adverse consequences, there are no interventions to meet the needs of these caregivers and their children. Resourcefulness Training, (cognitive-behavioral self-management intervention) has been shown to improve psychological and physical outcomes, mediate the effects of stress, and enhance the care provided to care-recipients. It will be tested in a randomized trial against an attention-only control arm. The intervention arm will receive an intervention that includes: a face-to-face session for teaching social (help-seeking) and personal (self-help) resourcefulness skills; ongoing access to video vignettes of caregivers of technology-dependent children describing resourcefulness skill application in daily life; 4 weeks of skills' reinforcement using daily journal writing; weekly phone calls for the first 4 weeks; and booster sessions at 2 and 4 months post enrollment. The Attention Control arm will receive weekly phone calls for the first 4 weeks and at 2 and 4 months post enrollment plus any usual care. The aims of the study are to: 1) Determine whether Resourcefulness Training versus Attention Control improves psychological (general mental health, depressive cognitions, depressive symptoms, appraised stress, burden) and physical outcomes (general physical health, chronic stress [hair cortisol]) and family functioning over 6 months in parents of technology-dependent children, after controlling for the parents' race/ethnicity, sex, family income, and children's functional status; and 2) Determine whether changes in psychological and physical outcomes and family functioning are mediated by changes in parents' levels of resourcefulness (personal and social). Data collection will take place at baseline then 6 weeks, 3 months, and 6 months post-enrollment. Our study will be the first to test a resourcefulness intervention for this caregiver population and to include male as well as female caregivers. This intervention is distinctive in that it uses web, telephone, and journal components for reinforcement-not multiple face-to-face visits that can be labor intensive. If shown to be efficacious, it can be easily replicated with other populations with strong potential for translation into practice.

ELIGIBILITY:
Inclusion Criteria:

* parent caregiver (biological, adoptive, or foster mother, father, grandmother or grandfather) for a technology-dependent child based on the Office of Technology Assessment (OTA) classification criteria (Group 1, mechanical ventilator; Group 2, intravenous nutrition/medication; Group 3 respiratory or nutritional support)
* at least 18 years of age
* able to speak and understand English due to the availability of the intervention and instruments in English only
* the technology-dependent child must be age 17 years or younger and receive care in the home from his/her parent

Exclusion Criteria:

* Parents of children with a cancer diagnosis will be excluded from participation due to the potentially life-threatening, terminal nature of the illness and grief reactions associated with a cancer diagnosis that may limit their ability to participate over the 6 month study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valerie A Toly, PhD, Principal Investigator — Frances Payne Bolton School of Nursing, Case Western Reserve University
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
The study team is still conducting analysis and writing up study results for publication.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Resourcefulness Training Intervention | Attention Control
Started | 46 | 47
Completed | 26 | 44
Not Completed | 20 | 3
Not completed — Lost to Follow-up | 5 | 3
Not completed — Protocol Violation | 4 | 0
Not completed — Withdrawal by Subject | 11 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Resourcefulness Training Intervention | Attention Control | Total
Number analyzed (Participants) | 46 | 47 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 45 | 90
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.5 (9.9) | 38.7 (10.8) | 39.1 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 40 | 78
  Male | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 43 | 44 | 87
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 14 | 24
  White | 30 | 28 | 58
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 46 | 47 | 93
General Physical Health [Mean (Full Range); unit: units on a scale] — Subjective Measure that is part of SF-12 survey that participants complete. The score range is 0-100, 0 indicates lowest level of health, 100 indicates highest level of health.
  units on a scale | 51.32 [27.33 to 67.74] | 49.48 [29.86 to 63.95] | 50.4 [27.33 to 67.74]
General Mental Health [Mean (Full Range); unit: units on a scale] — General Mental Health is a subjective survey that is part of the SF-12 Scale completed by participants. The score range is 0-100, 0 indicates lowest level of health, 100 indicates highest level of health.
  units on a scale | 42.6 [23.28 to 64.75] | 42.45 [17.48 to 60.68] | 42.5 [17.48 to 64.75]
Center for Epidemiological Studies- Depression [Mean (Full Range); unit: units on a scale] — This is commonly know as the CES-D. It is a subjective measure of depressive symptoms. Data is obtained via survey of participants. The score range is 0-60, Higher score indicates the presence of more symptomatology (more depressive symptoms).
  units on a scale | 19 [1 to 45] | 18.04 [1 to 41] | 18.5 [1 to 45]
Resourcefulness Scale [Mean (Full Range); unit: Score on a scale] — This subjective measure is collected via participant surveys. Score range is 0-140, higher score indicates greater resourcefulness.
  Score on a scale | 84.96 [51 to 129] | 87.52 [35 to 123] | 86.24 [35 to 129]
Depressive Cognitions Scale [Mean (Full Range); unit: units on a scale] — This is a subjective measure that is collected from participants via survey. Score range is 0-40, Higher Score indicates greater depressive cognition.
  units on a scale | 7.7 [0 to 28] | 8.4 [0 to 21] | 8.03 [0 to 28]
Feetham Family Functioning Survey [Mean (Standard Deviation); unit: units on a scale] — This subjective measure of family functioning is collected via participant survey. The score range is 0-175, which is the sum of the "differences" between reality and life expectations.
  Higher 'Difference' score indicates an imbalance between reality and life expectations
  units on a scale | 43.63 (29.39) | 39.57 (24.91) | 41.58 (27.14)
Zarit Burden Scale [Mean (Full Range); unit: units on a scale] — This is a subjective measure collected via participant survey. Score range is 0-48, higher score indicates greater burden.
  units on a scale | 20.1 [0 to 38] | 19.9 [2 to 39] | 20 [0 to 39]

OUTCOME MEASURES:

1. Primary Outcome: Depressive Cognitions Scale
Description: Subjective measure of participant depressive cognitions- precursor of depressive symptoms. Score range for the instrument is 0-40, where a higher score indicates greater depressive cognition.
Time Frame: From baseline to 6 weeks, 3 months, and 6 months post-enrollment
Measure: Mean (Full Range); unit: Score on a Scale
Arm/Group | Resourcefulness Training Intervention | Attention Control
Number analyzed (Participants) | 46 | 47
Score on a Scale
  6 Weeks Post Enrollment Timepoint | 6.46 [0 to 21] | 6.97 [0 to 26]
  3 Months Post Enrollment Timepoint | 6.32 [0 to 23] | 7.28 [0 to 32]
  6 Months Post Enrollment Timepoint | 5.65 [0 to 23] | 7.93 [0 to 40]

2. Primary Outcome: Medical Outcomes Short Form Health Survey (SF-12) Physical Health
Description: Change in General Mental and Physical Health from Baseline to 6 Months Post Enrollment. Score range is 0-100, where a '0' indicates lowest level of health, and '100' indicates highest level of health.
Time Frame: From baseline to 6 weeks, 3 months, and 6 months post-enrollment
Measure: Mean (Full Range); unit: Score on a Scale
Arm/Group | Resourcefulness Training Intervention | Attention Control
Number analyzed (Participants) | 46 | 47
Score on a Scale
  6 Weeks Post Enrollement Timepoint 2 | 52.7 [27 to 64.74] | 50.77 [28.26 to 66.51]
  3 Months Post Enrollment Timepoint 3 | 54.49 [28.39 to 67.02] | 49.46 [23.19 to 65.04]
  6 Months Post Enrollment Timepoint 4 | 51.49 [24.78 to 64.96] | 49.81 [24.43 to 62.29]

3. Primary Outcome: Medical Outcomes Short Form Health Survey (SF-12) Mental Health
Description: as for outcome 2
Time Frame: From baseline to 6 weeks, 3 months, and 6 months post-enrollment
Measure: Mean (Full Range); unit: Score on a Scale
Arm/Group | Resourcefulness Training Intervention | Attention Control
Number analyzed (Participants) | 46 | 47
Score on a Scale
  6 Weeks Post-Enrollment, Timepoint 2 | 47.02 [22.17 to 63.97] | 45.69 [17.8 to 61.42]
  3 Months Post-Enrollment, Timepoint 3 | 45.54 [26.17 to 63.5] | 47.41 [28.67 to 64.47]
  6 Weeks Post-Enrollment, Timepoint 4 | 49.51 [26.17 to 63.89] | 46.79 [15.15 to 62.05]

4. Secondary Outcome: Feetham Family Functioning Survey
Description: Change in Family Functioning from Baseline to 6 Months Post Enrollment. This subjective measure of family functioning is collected via participant survey. The score range is 0-175, which is the sum of the "differences" between reality and life expectations. Higher 'Difference' score indicates an imbalance between reality and life expectations
Time Frame: From baseline to 6 weeks, 3 months, and 6 months post-enrollment
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Resourcefulness Training Intervention | Attention Control
Number analyzed (Participants) | 46 | 47
Score on a Scale
  6 Weeks Post Enrollment Timepoint | 34.96 (22.01) | 36.38 (22.32)
  3 Months Post Enrollment Timepoint | 39.26 (22.83) | 37.44 (24.32)
  6 Months Post Enrollment Timepoint | 38.30 (23.66) | 32.43 (19.55)

5. Secondary Outcome: Resourcefulness Scale
Description: Subjective survey of participants' personal and social resourcefulness. Score range is 0-140, where a higher score indicates greater resourcefulness.
Time Frame: From baseline to 6 weeks, 3 months, and 6 months post-enrollment
Measure: Mean (Full Range); unit: Score on a Scale
Arm/Group | Resourcefulness Training Intervention | Attention Control
Number analyzed (Participants) | 46 | 47
Score on a Scale
  6 Weeks Post Enrollment Timepoint | 86.12 [50 to 125] | 93.59 [58 to 118]
  3 Months Post Enrollment Timepoint | 87.47 [60 to 102] | 88.22 [40 to 125]
  6 Months Post Enrollment Timepoint | 89.17 [22 to 121] | 93.59 [58 to 118]

ADVERSE EVENTS:
Time Frame: No adverse events were reported during the 6 month data collection period.
Description: The definitions do not differ in this context because no adverse events or serious adverse events were reported during the 6 month data collection period.
Arm/Group | Resourcefulness Training Intervention | Attention Control
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/46
Other Adverse Events (participants affected / at risk) | 0/46 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT03301831/Prot_SAP_004.pdf